CLINICAL TRIAL: NCT01390038
Title: Simpliciti IDE Trial
Brief Title: Simpliciti IDE Trial; Replacing the Humeral Head in Total Shoulder Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G100284
Record Dates: First submitted 2011-05-26; First posted 2011-07-08 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Primary Generalized (Osteo)Arthritis; Post-traumatic Arthrosis of Other Joints, Upper Arm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Simpliciti™ Shoulder System (Experimental): The Simpliciti™ Shoulder System is intended for Total Shoulder Arthroplasty of the shoulder.
  Interventions: Device: Simpliciti™ Shoulder System

INTERVENTIONS:
Device: Simpliciti™ Shoulder System — Total shoulder arthroplasty system

SUMMARY:
The purpose of this study is to demonstrate safety and efficacy of the Simpliciti Shoulder System in total shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject 22 years or older
* Clinical indication for total shoulder replacement due to primary diagnosis of arthritis. Primary arthritis for this study includes osteoarthritis, and/or traumatic arthritis.
* Scapula and proximal humerus must have reached skeletal maturity
* Subject with a Constant Score ≥ 20
* Willing and able to comply with the protocol
* Willing and able to sign the informed consent (or the Legally Authorized Representative will sign for the subject)

Exclusion Criteria:

* Lack of sufficient sound bone to seat and support the implant such as:

  1. Rapid joint destruction, marked bone loss or bone resorption;
  2. Destruction of the proximal humerus that precludes rigid fixation of the humeral component; and
  3. Osteomalacia
* Metal allergies or sensitivity, including a known allergic reaction to implant metals (e.g., nickel) or polyethylene
* Infection at or near the site of implantation, including:

  1. Glenohumeral joint infection
  2. Osteomyelitis
* Distant or systemic infection
* Medical conditions or balance impairments that could lead to falls
* Prior open shoulder surgery on the shoulder to be treated in the study including failed rotator cuff surgery, but excluding successful shoulder arthroscopy
* Any full thickness rotator cuff tear at the time of surgery or a nonfunctional rotator cuff
* Excessive glenoid bone loss defined by preoperative computed tomography (CT) scans of the shoulder which show insufficient glenoid bone, or insufficient bone identified at the time of surgery
* Metabolic disorders which may impair bone function
* Nonfunctional deltoid muscle
* Neuromuscular compromise condition of the shoulder (e.g., neuropathic joints or brachioplexus injury with a flail shoulder joint)
* Known active metastatic or neoplastic diseases, Paget's disease or Charcot's disease
* Currently, or within the last 6 months, or planning to be on chemotherapy or radiation
* Currently taking > 5mg/day corticosteroids (e.g. prednisone) excluding inhalers, within 3 months prior to surgery
* Female subjects who are pregnant or planning to become pregnant within the study period
* In the surgeon's opinion, the subject is unable to understand the study or be compliant with the follow up or have a history of non-compliance with medical advice
* History of any cognitive or mental health status that would interfere with study participation
* Alcohol or drug abuse
* Engages in manual labor or sports activities that could affect shoulder outcome
* Currently enrolled in any clinical research study that might interfere with the current study endpoints

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2011-07; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Saint Agnes Medical Center, Fresno, California
  - Grossmont/Sharp Hospital, La Mesa, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Rush Hospital, Chicago, Illinois
  - Beverly Hills Orthopaedic Surgery, Beverly Hills, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Sports and Orthopaedic Specialists, Edina, Minnesota
  - University of Missouri-Columbia, Columbia, Missouri
  - Bassett Healthcare Network Research Institute, Cooperstown, New York
  - Cleveland Clinic, Euclid, Ohio
  - The Center, Bend, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Knoxville Orthopaedic Clinic, Knoxville, Tennessee
  - Aurora Medical Center - Grafton, Grafton, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Simpliciti™ Shoulder System
Started | 157
Completed | 149
Not Completed | 8
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 4
Not completed — Simpliciti System Removal | 2

BASELINE CHARACTERISTICS:
Arm/Group | Simpliciti™ Shoulder System
Number analyzed (Participants) | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 112

OUTCOME MEASURES:

1. Primary Outcome: Device Success Rate
Description: A subject is a Patient Success at 24-months if:
  1. There is NO continuous radiolucent line around the prosthesis; and
  2. The adjusted Constant Score is > 85 (successful outcome); and
  3. They did not have revision surgery; and
  4. They did not have a system-related serious adverse event.
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Simpliciti™ Shoulder System
Number analyzed (Participants) | 149
participants | 134

2. Secondary Outcome: Quality of Life
Description: Simple Shoulder Test
  1 (worse) - 12 (best)
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Simpliciti™ Shoulder System
Number analyzed (Participants) | 148
units on a scale | 10.8 (1.7)

3. Secondary Outcome: Range of Motion
Description: * Elevation in the scapula plane
  * Internal rotation with arm at the side
  * External rotation with arm at the side
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Simpliciti™ Shoulder System
Number analyzed (Participants) | 149
Degrees
  Elevation in the Scapular Plan | 146.6 (23.7)
  Internal Rotation | 73.9 (1635)
  External Rotation | 56.4 (15.4)

4. Secondary Outcome: Strength
Description: Strength of a Specific shoulder motion as measured in pounds of force on a dynamometer machine supplied by Tornier
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Simpliciti™ Shoulder System
Number analyzed (Participants) | 143
Pounds | 15.7 (7.8)

5. Secondary Outcome: Device Parameters
Description: Devices will be assessed to determine percentage of participants that demonstrated the following after total shoulder arthroplasty:
  * Migration
  * Osteolysis
  * Subsidence
Time Frame: 24 months
Measure: Number; unit: Percentage of participants
Arm/Group | Simpliciti™ Shoulder System
Number analyzed (Participants) | 149
Percentage of participants
  Migration | 0
  Osteolysis | 0
  Subsidence | 0

6. Secondary Outcome: American Shoulder and Elbow Surgeon Score
Description: 0 (worst) - 100 (best)
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Simpliciti™ Shoulder System
Number analyzed (Participants) | 149
units on a scale | 91.9 (11.4)

7. Secondary Outcome: Pain: Visual Analog Scale
Description: 0 (best) - 10 (worst)
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Simpliciti™ Shoulder System
Number analyzed (Participants) | 149
units on a scale | 0.5 (1.2)

ADVERSE EVENTS:
Arm/Group | Simpliciti™ Shoulder System
Serious Adverse Events (participants affected / at risk) | 4/157
Other Adverse Events (participants affected / at risk) | 51/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simpliciti™ Shoulder System (N=157)
Aseptic Glenoid Loosening (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthrofibrosis, treated shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simpliciti™ Shoulder System (N=157)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 39 (46) — OA in other joints leading to joint replacement
Pain (Musculoskeletal and connective tissue disorders) | 12 (13) — Not related to the study shoulder

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs are restricted from publishing study results until either 18 months after the study is completed or the primary manuscript has been accepted, whichever comes first.